CLINICAL TRIAL: NCT05924243
Title: A Phase 1b, Adaptive, Multi-Center, Randomized, Double Blind, Placebo-Controlled, Parallel Design Study to Investigate The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7486967 in Participants With Early Idiopathic Parkinson's Disease
Brief Title: A Study to Investigate The Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO7486967 in Participants With Early Idiopathic Parkinson's Disease.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BP43176
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RO7486967 Arm (Experimental): Participants will receive RO07486967 for approximately 28 days with 14 days of follow up after the last dose.
  Interventions: Drug: RO7486967
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RO7486967 — For up to approximately 28 days
  Arms: RO7486967 Arm
Drug: Placebo — For up to approximately 28 days
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, adaptive, parallel-group, placebo controlled Phase 1b study to evaluate the safety, tolerability, pharmacokinetic (PK) and pharmacodynamics of RO7486967 in participants with idiopathic PD at the early stage of the disease (modified H&Y stage ≤2.5) who are either treatment-naïve or on stable treatment with symptomatic therapy (levodopa and/or pramipexole, ropinirole, rotigotine).

ELIGIBILITY:
Inclusion Key Criteria:

* Male or post-menopausal female
* Diagnosis of clinically probable idiopathic PD based on MDS criteria with bradykinesia plus one of the other cardinal signs of PD (resting tremor, rigidity)
* A time from diagnosis of PD of at least 3 to maximum 60 months (5 years) at screening
* Modified H&Y Stage ≤2.5 (in ON state)
* Dopaminergic imaging consistent with dopamine transporter deficit
* "High-affinity binder" or "mixed-affinity binder" genotype for TSPO
* Either treatment naïve or treatment with symptomatic PD therapy (levodopa and/or pramipexole, ropinirole, rotigotine) given for at least 90 days, with stable doses for at least 30 days prior to the first dose
* No anticipated changes in PD therapy throughout the study duration
* SARS-CoV-2 vaccination completed at least 60 days prior to the first dose.

Exclusion Key Criteria:

* Medical history indicating a Parkinsonian syndrome other than idiopathic PD
* CNS or psychiatric disorders other than idiopathic PD (mild depression or anxiety arising in the context of PD is not exclusionary)
* History of brain surgery for PD
* Use of any of symptomatic drug for PD other than levodopa pramipexole, ropinirole, or rotigotine within 60 days prior to the first dose
* Known carriers for mutations in the following genes: alpha-synuclein, LRRK2, GBA, PRKN, PINK1, or DJ1
* Unstable or clinically significant cardiovascular disease within the last year prior to screening
* Uncontrolled hypertension
* Use of oral anticoagulants, low-molecular-weight heparin, warfarin (Coumadin), acenocoumarol, and phenprocoumon is not allowed within 10 days before the first Lumbar Puncture and during the study (low dose aspirin is permitted as monotherapy)
* Concomitant disease or unstable medical condition within 6 months of screening that could interfere with the study or treatment that might interfere with the conduct of the study, including but not limited to autoimmune disease, immunodeficiency diseases, any active infectious disease
* History of immunodeficiency diseases
* Presence of hepatitis B surface antigen (HBsAg) or positive for total hepatitis B core antibody (HBcAb), or positive hepatitis C (HCV) at screening
* Vaccine(s) other than SARS-CoV2 vaccine within 28 days prior to the first dose, or plans to receive vaccines during the study or within 28 days of the last dose
* History of chronic liver disease
* Clinically significant abnormalities in laboratory test results at screening, including hepatic and renal panels, complete blood count, chemistry panel and urinalysis
* Any previous administration of RO7486967 or other compound targeting NLRP3
* Enrollment in another investigational study
* Use of any of other investigational therapy (other than protocol-mandated study treatment) within 90 days or 5 drug elimination half-lives (whichever is longer) prior to the first dose

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-07-18 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with adverse events (AEs) | Up to 45 Days
The change in Columbia-Suicide Severity Rating Scale (C-SSRS) Scores from baseline | From Baseline to Up to 45 Days

SECONDARY OUTCOMES:
Time to maximum concentration of RO7486967 in Plasma | Day 1, Day 15, and Day 28
Maximum concentration (Cmax) of RO7486967 in Plasma | Day 1, Day 15, and Day 28
Area under the curve (AUC) RO7486967 in Plasma | Day 1, Day 15, and Day 28
Change from baseline in parametric bindings of [18F]-DPA-714 in different brain areas at Day 25 PET | From Baseline to Approximately Day 25

CONTACTS AND LOCATIONS:
Locations (17):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Cedars Sinai Medical Center, Los Angeles, California
  - CenExel Rocky Mountain Clinical Research, LLC, Englewood, Colorado
  - Georgetown University, Washington D.C., District of Columbia
  - Advent Health Orlando, Orlando, Florida
  - Quest Research Institute, Farmington Hills, Michigan
  - Weill Cornell Medical College, New York, New York
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - University Pennsylvania Hospital, Philadelphia, Pennsylvania
- Netherlands (3):
  - Brain Research Center B.V, Amsterdam
  - UMC St Radboud, Nijmegen
  - Brain Research Center Zwolle, Zwolle
- United Kingdom (5):
  - University of Exeter, Exeter
  - Barts Health NHS Trust, London
  - Imperial College Healthcare NHS Trust; Charing Cross Hospital, London
  - National Hospital for Neurology and Neurosurgery; Leonard Wolfson Experimental Neurology Centre CRF, London
  - Campus for Ageing & Vitality; Clincal Ageing Research Unit, Newcastle

IPD SHARING:
Plan to Share IPD: No
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).